CLINICAL TRIAL: NCT02624921
Title: Positive Health Effects of the Natural Outdoor Environment in Typical Populations in Different Regions in Europe. Work Package 4: Therapeutic Study in Barcelona
Brief Title: PHENOTYPE. Therapeutic Study in Barcelona
Status: Completed | Type: Observational
Sponsor: Barcelona Institute for Global Health (Other)
Responsible Party: Principal Investigator, Mark Nieuwenhuijsen, Air Pollution and Urban Environment program coordinator, Barcelona Institute for Global Health
Other Study IDs: PHENOTYPE_WP4BCN
Record Dates: First submitted 2015-12-01; First posted 2015-12-09 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Poor Mental Health; Natural Outdoor Environments

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

INTERVENTIONS:
Other: There was no intervention. — Participants were transported one day to a urban setting, one day to a green space, one day to a beach. No intervention was done.

SUMMARY:
The study aimed to explore therapeutic effects of natural environments. To do so, the investigators evaluated the immediate and sustained changes in several indicators of well-being while people (n=26) with poor mental health were engaged in unconstrained exposures to natural (green, blue) and urban environments. The indicators included: affection, cognition, physiological responses.

Each participant was exposed to all environments for a period of 210 minutes between October 2013 and January 2014. During the exposure period, participants were instructed to do what they would usually do in that environment. Before, during (at 30 and 210 minutes) and after each exposure, several psycho-physiological measures were taken: (i) heart rate variability and heart rate using a Holter monitor, (ii) blood pressure using a digital blood pressure monitor, (iii) physical activity using the CalFIT application installed in a Smartphone, (iv) lung function using a portable computerized spirometer, (v) stress level using salivary cortisol samples collected using Salivettes, (vi) affect, perceived restoration and social interactions using questionnaires, (vii) cognitive functioning using the backwards digit-span task test.

ELIGIBILITY:
Inclusion Criteria:

* MHI-5 scored in the lower 50th percentile of the Barcelona city PHENOTYPE sample
* willing to participate

Exclusion Criteria:

* no able to walk for 30 minutes at self-directed pace.
* with chest, abdomen surgery or heart attack during the last three months.
* with retinal detachment or eyes surgery or hospitalized for heart problem during the last month.
* with tuberculosis treatment, or respiratory infection during the last three weeks.
* being asthmatic or pregnant
* using inhaler the 24 hours previous to the study day.
* taking medication different from the usual the 24 hours previous to the study day.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the participants (n=26) were individuals that had previously participated in a survey of 1000 people in Barcelona city as part of the PHENOTYPE project. As part of the survey, they had answered the Mental Health Inventory (MHI-5) subscale from the SF-36 health questionnaire. The investigators purposively selected those individuals MHI-5 scored in the lower 50th percentile.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline heart rate variability at 30 min | after 30 minutes of exposure to green/blue/urban environment
Change from Baseline heart rate at 30 min | after 30 minutes of exposure to green/blue/urban environment
Change from blood pressure at 30min | after 30 minutes of exposure to green/blue/urban environment
Change from stress level at 30min (salivary cortisol) | after 30 of exposure to green/blue/urban environment
Change from affect at 30 min (BRUMS/POMS) | after 30 minutes of exposure to green/blue/urban environment
Change from cognitive functioning at 30 min (backward digit span task) | after 30 minutes of exposure to green/blue/urban environment
Change from Baseline heart rate variability at 210 min | after 210 minutes of exposure to green/blue/urban environment
Change from Baseline heart rate at 210 min | after 210 minutes of exposure to green/blue/urban environment
Change from blood pressure at 210min | after 210 minutes of exposure to green/blue/urban environment
Change from stress level at 210min (salivary cortisol) | after 210 minutes of exposure to green/blue/urban environment
Change from affect at 210 min (BRUMS/POMS) | after 210 minutes of exposure to green/blue/urban environment
Change from cognitive functioning at 210 min (backward digit span task) | after 210 minutes of exposure to green/blue/urban environment

SECONDARY OUTCOMES:
objectively measured physical activity 30 | During the first 30 minutes of exposure to green/blue/urban environment
  Measured with a Smartphone application (CalFIT)
perceived restoration 30 (ROS - Korpela's Restoration outcome scale) | after 30 minutes of exposure to green/blue/urban environment
subjectively recorded social interactions 30 | after 30 minutes of exposure to green/blue/urban environment
  Measurement tool developed by the research team
ambient air pollution exposure 30 (PM2.5) | During the first 30 minutes of exposure to green/blue/urban environment
  Measured with MicroAthelometer
objectively measured physical activity 210 | During the first 210 minutes of exposure to green/blue/urban environment
  Measured with a Smartphone application (CalFIT)
perceived restoration 210 (ROS- Korpela's Restoration outcome scale) | after 210 minutes of exposure to green/blue/urban environment
subjectively recorded social interactions 210 | after 210 minutes of exposure to green/blue/urban environment
  Measurement tool developed by the research team
ambient air pollution exposure 210 (PM2.5) | During the first 210 minutes of exposure to green/blue/urban environment
  Measured with MicroAthelometer
personal air pollution (CO, NO, NO2) | During all the data collection day
  Personal sensors designed and built at Cambridge University, UK (CamPerS)

REFERENCES:
- [Derived] Triguero-Mas M, Gidlow CJ, Martinez D, de Bont J, Carrasco-Turigas G, Martinez-Iniguez T, Hurst G, Masterson D, Donaire-Gonzalez D, Seto E, Jones MV, Nieuwenhuijsen MJ. The effect of randomised exposure to different types of natural outdoor environments compared to exposure to an urban environment on people with indications of psychological distress in Catalonia. PLoS One. 2017 Mar 1;12(3):e0172200. doi: 10.1371/journal.pone.0172200. eCollection 2017. PMID 28248974